CLINICAL TRIAL: NCT04000672
Title: Patient Specific Instrumentation (PSI) Referencing Osteotomy Technological Transfer and Education - a PSI High Tibial Osteotomy, Double-blinded, Randomized Controlled Trial - the PROTECTED HTO (High Tibial Osteotomy) Trial
Brief Title: Patient Specific Instrumentation (PSI) Referencing Osteotomy Technological Transfer - a Randomized Control Trial (RCT)
Acronym: ProtectedHTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lawrence CM Lau, Principle Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019.050
Record Dates: First submitted 2019-06-22; First posted 2019-06-27 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Osteotomy; Randomized Controlled Trial
Keywords: Patient Specific Instrumentation; Randomized controlled trial; High Tibial Osteotomy

STUDY DESIGN:
Intervention Model Description: Control group: High tibial osteotomy with navigation Intervention group: High tibial osteotomy with navigation and PSI jig
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be accomplished by computer-generated randomization sequence using serially numbered opaque, sealed envelopes with patients assigned either to intervention or control groups. All investigators, research staff, patients except the surgeon performing the HTO will be blinded to the group assignment of the subjects. Nor they will be aware of the regimen prescribed during the study and evaluation periods. A randomization code will be allocated to each included subjects to maintain blindness. Randomization code will be broken only after the database had been locked. Patient rehabilitation, post-operative assessment and Data analysis are conducted by personnel blinded to the patients' randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTO with navigation (Active Comparator): High Tibial Osteotomy is offered to patients with symptomatic medial compartment knee osteoarthritis (OA)
  Interventions: Procedure: HTO with navigation
- HTO with navigation + PSI jig (Experimental): 3D printed patient specific metal jigs (PSI jig) are created based on the pre-operative CT image. After that, calibrated osteotome is used to achieve the desired correction with the use of navigation for overall lower limb alignment, which is the same as the "Active Comparator" group.
  Interventions: Procedure: 3D printed patient specific metal jigs (PSI jig); Procedure: HTO with navigation

INTERVENTIONS:
Procedure: 3D printed patient specific metal jigs (PSI jig) — PSI jig is created based on the pre-operative CT image. Standard medial open wedge osteotomy described previously is performed. Incision is made in the midway between posteromedial border of the tibia and medial aspect of the tibial tuberosity. Sartorius fascia is cut and retracted medially to expose the medial collateral ligament (MCL). Then the PSI jig is positioned onto the tibia. Due to the jig patient specific design (individually based on each patient's CT image), it can fit closely to the proximal tibia. The slot opening on the PSI jig corresponds to 4 cm below the medial joint line and the slot design allow the sawblade cut direction toward the safe zone of the lateral cortex under fluoroscopy. The PSI Jig is removed after the bone cut completed and would not retain in patient's body.
  Arms: HTO with navigation + PSI jig
Procedure: HTO with navigation — In brief, an incision is made in the midway between posteromedial border of the tibia and medial aspect of the tibial tuberosity. Sartorius fascia is cut and retracted medially to expose the medial collateral ligament (MCL). Two to three K-wires are placed 4 cm below the medial joint line toward the safe zone (an area between the tip of the fibular head and the remnant of fibular head epiphysis line) of the lateral cortex under fluoroscopy and osteotomy is done below and parallel to the k-wires using an oscillating saw leaving the lateral 10 mm intact.

SUMMARY:
Medial open wedge high tibial osteotomy is a surgery performed to treat knee osteoarthritis in young patients.Recently with our department advance of technology, the investigators performed computed tomography for the patient's lower limb and 3D reconstruct the image. Based on the 3D image, the investigators planned our planned osteotomy cut on computer software Materialize 3 and the investigators then 3D printed a metal jig that has a slot to produce the osteotomy and also protected the neurovascular bundles. Therefore these metal jigs are specific to each patients. The investigators have performed a few cases of HTO under this extra metal jig protection and guidance and noted it has improved accuracy and safety clinically. However, whether it has scientific significance difference in accuracy is not known.

DETAILED DESCRIPTION:
Medial open wedge high tibial osteotomy is a surgery performed to treat knee osteoarthritis in young patients. Currently the investigators perform high tibial osteotomy under the guidance of computer navigation to achieve the required alignment. During conventional high tibial osteotomy the bone cut is done by free hand cutting, there are risks of cutting into the posterior proximal tibia compartment and transect the neurovascular bundles which is a surgical disaster and may then lead to loss of limb. And the accuracy of free hand cutting is limited by experience of surgeons. In our conventional high tibial osteotomy transection of neurovascular bundles has never happened given our meticulous surgical technique but the investigators believe an extra protection is always beneficial to our patients. Recently with our department advance of technology, the investigators performed computed tomography for the patient's lower limb and 3D reconstruct the image. Based on the 3D image, the investigators planned our planned osteotomy cut on computer software Materialize 3 and the investigators then 3D printed a metal jig that has a slot to produce the osteotomy and also protected the neurovascular bundles. Therefore these metal jigs are specific to each patients. The investigators have performed a few cases of HTO under this extra metal jig protection and guidance and noted it has improved accuracy and safety clinically. However, whether it has scientific significance difference in accuracy is not known.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patient with medial compartment knee OA
* medial compartment OA was grade 3 or milder according to Kellgren-Lawrence classification

Exclusion Criteria:

* lateral compartment OA
* symptomatic patellofemoral compartment OA,
* inflammatory arthritis,
* significant loss of knee joint range in flexion (less than 100°) or in extension (less than - 10°),
* ligamentous instability,
* obesity with a body mass index greater than 30,
* significant psychological disorder
* inability to communicate in Chinese or English language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Knee Society knee score | 1 week before surgery
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Knee Society knee score | 6 months post-op
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Knee Society knee score | 1 year post-op
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Knee Society knee score | 2 year post-op
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Knee Society function score | 1 week before surgery
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Knee Society function score | 6 months post-op
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Knee Society function score | 1 year post-op
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Knee Society function score | 2 year post-op
  Clinical and functional scores, on a 100-point scale; Knee Society score (KSS) has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. "Excellent" for score 80-100, "Good" for score 70-79, "Fair" for score 60-69, "Poor" for score below 60.
Oxford Knee Score | 1 week before surgery
  Clinical and functional scores
Oxford Knee Score | 6 months post-op
  Clinical and functional scores
Oxford Knee Score | 1 year post-op
  Clinical and functional scores
Oxford Knee Score | 2 year post-op
  Clinical and functional scores
Range of motion | 1 week before surgery
  Evaluated using a manual goniometer
Range of motion | 1 week before discharge
  Evaluated using a manual goniometer
Range of motion | 3 months post-op
  Evaluated using a manual goniometer
Range of motion | 6 months post-op
  Evaluated using a manual goniometer
Range of motion | 1 year post-op
  Evaluated using a manual goniometer
Range of motion | 2 year post-op
  Evaluated using a manual goniometer
Pain Visual Analog Scale (VAS) score | 1 week before surgery
  The VAS is a psychometric response scale and a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The VAS pain ranges 0-10, with 10 representing the most pain.
Pain Visual Analog Scale (VAS) score | 1 week before discharge
  The VAS is a psychometric response scale and a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The VAS pain ranges 0-10, with 10 representing the most pain.
Pain Visual Analog Scale (VAS) score | 3 months post-op
  The VAS is a psychometric response scale and a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The VAS pain ranges 0-10, with 10 representing the most pain.
Pain Visual Analog Scale (VAS) score | 6 months post-op
  The VAS is a psychometric response scale and a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The VAS pain ranges 0-10, with 10 representing the most pain.
Pain Visual Analog Scale (VAS) score | 1 year post-op
  The VAS is a psychometric response scale and a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The VAS pain ranges 0-10, with 10 representing the most pain.
Pain Visual Analog Scale (VAS) score | 2 year post-op
  The VAS is a psychometric response scale and a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. The VAS pain ranges 0-10, with 10 representing the most pain.
Measurement of knee displacement | 1 week before surgery
  Measure the displacement (in cm) between femoral head and tibial head on a secured computer using CT scan images and scanogram images
Measurement of knee displacement | 1 year after surgery
  Measure the displacement (in cm) between femoral head and tibial head on a secured computer using CT scan images and scanogram images

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital & Alice Ho Miu Ling Nethersole Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data and resources will be shared with other eligible investigators through academically established means. The protocol and datasets used and/or analysed in this study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after study completes
Access Criteria: Data and resources will be shared with other eligible investigators through academically established means. The protocol and datasets used and/or analysed in this study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Lau LCM, Chui ECS, Fan JCH, Man GCW, Hung YW, Ho KKW, Chung KY, Wan SYC, Chau JWW, Yung PSH, Bhandari M. Patient-specific instrumentation (PSI) Referencing High Tibial Osteotomy Technological Transfer and Education: protocol for a double-blind, randomised controlled trial (PROTECTED HTO Trial). BMJ Open. 2021 Feb 5;11(2):e041129. doi: 10.1136/bmjopen-2020-041129. PMID 33550239